CLINICAL TRIAL: NCT00958711
Title: The Mechanism of Action of the Unite Biomatrix in Diabetic Foot Ulcer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Budgetary
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Synovis Surgical Innovations (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U-0801
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biologic - Unite Biomatrix (Experimental)
  Interventions: Device: Unite Biomatrix
- Saline and Gauze (Active Comparator)
  Interventions: Other: Saline and Gauze

INTERVENTIONS:
Device: Unite Biomatrix — Collagen based, decellularized equine pericardial dressing for skin surface wounds
  Arms: Biologic - Unite Biomatrix
Other: Saline and Gauze — gauze moistened with sterile saline
  Arms: Saline and Gauze

SUMMARY:
The purpose of this study is to assess the mechanism of action of the Unite Biomatrix and compare its performance with the standard of care, saline moistened gauze, for the treatment of diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. A full thickness diabetic foot ulcer with a viable wound bed free of necrotic material (grade 1 on Wagner scale).
2. Diagnosis of diabetes mellitus (type I or II) adequately controlled.
3. The ulcer is greater than 4 weeks duration.
4. Three or fewer ulcers separated by > 3.0 cm distance.
5. Post-debridement, the ulcer size must be between 1 and 10 sq cm2.
6. Ankle/brachial index is between 0.7 to 1.2 and or one of the following must be present:

   * transcutaneous partial pressure oxygen (TcPO2) > 30 mmHg at the ankle
   * toe pressure of >40mm Hg or a Doppler waveform consistent with adequate flow in the foot (biphasic or triphasic)
7. At least 18 years old.
8. Able and willing to provide a voluntary written informed consent.
9. Able and willing to wear an off-loading orthopedic shoe.
10. Able and willing to attend scheduled follow-up visits and study related exams.

Exclusion Criteria:

1. Greater than 30% reduction in wound size during first week of observation by the investigator.
2. Ulcer with exposed tendon or bone.
3. Gross clinical infection at the study ulcer site including cellulitis and osteomyelitis.
4. Gangrene.
5. Active Charcot's disease as determined by clinical and radiographic examination.
6. Ulcer of a non-diabetic pathophysiology (e.g., rheumatoid, radiation-related, and vasculitis related ulcers).
7. Known severe anemia.
8. Known serum albumin < 2.5.
9. Renal failure with Creatinine > 2.5.
10. Rheumatoid arthritis (and other collagen vascular disease), vasculitis, sickle cell disease, HIV.
11. Severe liver disease as defined by the treating physician or patient's primary care physician.
12. Malignancy at or near the ulcer site.
13. Any condition judged by the investigator that would cause the study to be detrimental to the patient.
14. Presence of a hematology, clinical, chemistry or other test obtained within 7 days of screening that is outside the normal range for the laboratory and is determined to be clinically significant by the investigator.
15. Received another investigational device or drug within 30 days of Day 0.
16. Radiation therapy, chemotherapy or immunosuppressive therapy within 30 days of enrollment.
17. Received another allograft, autograft or xenograft within 30 days of the Day 0.
18. Known allergy to equine derived tissue.
19. Alcohol or drug abuse, defined as current medical treatment for substance abuse.
20. Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of California - San Diego, San Diego, California
  - University of Miami, Miller School of Medicine, Miami, Florida
  - Aiyan Diabetes Center, Evans, Georgia
  - Foot & Ankle Associates of Central Illinois, LLC, Springfield, Illinois
  - Eastern Carolina Foot and Ankle, Greenville, North Carolina
  - Foot and Ankle East, Greenville, North Carolina
  - Carolina East Family Medicine, Greenville, North Carolina
  - Family Foot & Ankle Physicians, Greenville, North Carolina
  - Comprehensive Wound Care Thoracic & Vascular Associates of Kinston P.A., Kinston, North Carolina
  - The Foot & Ankle Associates of North Carolina, PLLC, Rocky Mount, North Carolina
  - Martin Foot and Ankle, York, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Biologic - Unite Biomatrix | Saline and Gauze
Started | 42 | 48
Completed | 29 | 27
Not Completed | 13 | 21
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Physician Decision | 5 | 7
Not completed — Lost to Follow-up | 4 | 1
Not completed — Other | 2 | 5
Not completed — Death | 1 | 2
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biologic - Unite Biomatrix | Saline and Gauze | Total
Number analyzed (Participants) | 42 | 48 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (10.7) | 54.9 (10.2) | 56.39 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 32 | 34 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 24 | 24 | 48
  Black | 11 | 19 | 30
  Hispanic | 6 | 4 | 10
  Pacific Islander | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Not Healed by Number of Days After Procedure
Description: Time to complete healing was captured by Kaplan-Meier Plot showing percentage of participants not healed by number of days after procedure. Patients were considered healed at their first follow-up visit where the patient's would had healed.
Time Frame: Day 20, Day 40, Day 60, Day 80
Population: Intent-to-Treat (ITT): all randomized participants who provided consent..
Measure: Number; unit: Percentage of Participants
Arm/Group | Biologic - Unite Biomatrix | Saline and Gauze
Number analyzed (Participants) | 42 | 48
Percentage of Participants
  Day 20 | 0.97 | 1.0
  Day 40 | 0.91 | 0.95
  Day 60 | 0.74 | 0.74
  Day 80 | 0.61 | 0.65

2. Primary Outcome: Percentage of Participants With Wounds Healed at 12 Weeks
Time Frame: Week 12
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Biologic - Unite Biomatrix | Saline and Gauze
Number analyzed (Participants) | 42 | 48
Percentage of participants
  Healed | 42.9 | 29.2
  Not Healed | 57.1 | 70.8

3. Primary Outcome: Wound Healing Pathway Markers
Time Frame: Day 0, 72 hours post-procedure, Week 1, Week 2, Week 4
Population: Source document notes "no data provided." Limited information available since product no longer licensed with Baxter.
Arm/Group | Biologic - Unite Biomatrix | Saline and Gauze
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Bacterial Burden
Time Frame: Day 0, Week 1 - Week 12
Population: Source document notes "no data provided." Limited information available since product no longer licensed with Baxter.
Arm/Group | Biologic - Unite Biomatrix | Saline and Gauze
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage Mean of Original Wound Size From Baseline by Week
Description: The percent of original wound size was calculated using the following formula: measure at baseline minus measure at follow-up visit divided by measure at baseline. In cases when the baseline depth was reported as 0cm, the minimum non-zero value in the sample (0.1cm) was imputed so a percent reduction measure could be calculated.
Time Frame: Day 0, Week 4, Week 8, Week 12
Population: ITT
Measure: Mean (Standard Deviation); unit: Percentage mean of wound size
Arm/Group | Biologic - Unite Biomatrix | Saline and Gauze
Number analyzed (Participants) | 42 | 48
Percentage mean of wound size
  Week 4 Length: number analyzed (Participants) | 35 | 39
  Week 4 Length | 0.879 (NA) — Study sponsored by other company, and only abbreviated results available without this data point. | 0.754 (NA) — Study sponsored by other company, and only abbreviated results available without this data point.
  Week 4 Width: number analyzed (Participants) | 35 | 39
  Week 4 Width | 0.809 (NA) — Study sponsored by other company, and only abbreviated results available without this data point. | 0.750 (NA) — Study sponsored by other company, and only abbreviated results available without this data point.
  Week 4 Depth: number analyzed (Participants) | 22 | 40
  Week 4 Depth | 0.820 (NA) — Study sponsored by other company, and only abbreviated results available without this data point. | 1.082 (NA) — Study sponsored by other company, and only abbreviated results available without this data point.
  Week 4 Area: number analyzed (Participants) | 36 | 39
  Week 4 Area | 0.807 (NA) — Study sponsored by other company, and only abbreviated results available without this data point. | 0.732 (NA) — Study sponsored by other company, and only abbreviated results available without this data point.
  Week 8 Length: number analyzed (Participants) | 22 | 28
  Week 8 Length | 0.705 (NA) — Study sponsored by other company, and only abbreviated results available without this data point. | 0.695 (NA) — Study sponsored by other company, and only abbreviated results available without this data point.
  Week 8 Width: number analyzed (Participants) | 22 | 28
  Week 8 Width | 0.650 (NA) — Study sponsored by other company, and only abbreviated results available without this data point. | 0.671 (NA) — Study sponsored by other company, and only abbreviated results available without this data point.
  Week 8 Depth: number analyzed (Participants) | 10 | 28
  Week 8 Depth | 1.612 (NA) — Study sponsored by other company, and only abbreviated results available without this data point. | 1.365 (NA) — Study sponsored by other company, and only abbreviated results available without this data point.
  Week 8 Area: number analyzed (Participants) | 23 | 28
  Week 8 Area | 0.546 (NA) — Study sponsored by other company, and only abbreviated results available without this data point. | 0.592 (NA) — Study sponsored by other company, and only abbreviated results available without this data point.
  Week 12 Length: number analyzed (Participants) | 24 | 26
  Week 12 Length | 0.381 (NA) — Study sponsored by other company, and only abbreviated results available without this data point. | 0.567 (NA) — Study sponsored by other company, and only abbreviated results available without this data point.
  Week 12 Width: number analyzed (Participants) | 24 | 26
  Week 12 Width | 0.323 (NA) — Study sponsored by other company, and only abbreviated results available without this data point. | 0.465 (NA) — Study sponsored by other company, and only abbreviated results available without this data point.
  Week 12 Depth: number analyzed (Participants) | 16 | 26
  Week 12 Depth | 0.304 (NA) — Study sponsored by other company, and only abbreviated results available without this data point. | 1.347 (NA) — Study sponsored by other company, and only abbreviated results available without this data point.
  Week 12 Area: number analyzed (Participants) | 25 | 26
  Week 12 Area | 0.341 (NA) — Study sponsored by other company, and only abbreviated results available without this data point. | 0.433 (NA) — Study sponsored by other company, and only abbreviated results available without this data point.

6. Secondary Outcome: Number of Participants With Ulcer Recurrence
Time Frame: Week 1 to Week 24
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Biologic - Unite Biomatrix | Saline and Gauze
Number analyzed (Participants) | 42 | 48
Participants | 0 | 2

7. Secondary Outcome: Number of Device-related Adverse Events (AE)
Time Frame: Week 1 to Week 24
Population: ITT
Measure: Number; unit: Events
Arm/Group | Biologic - Unite Biomatrix | Saline and Gauze
Number analyzed (Participants) | 42 | 48
Events | 0 | 0

8. Secondary Outcome: Number of Procedure-related Adverse Events (AE)
Time Frame: Week 1 to Week 24
Population: ITT
Measure: Number; unit: Events
Arm/Group | Biologic - Unite Biomatrix | Saline and Gauze
Number analyzed (Participants) | 42 | 48
Events | 2 | 0

9. Secondary Outcome: Number of Device Failures
Description: Includes failure to heal the ulcer by the 12-week visit under the Intent-to-Treat principle.
Time Frame: Week 1 to Week 24
Population: ITT
Measure: Number; unit: Devices
Arm/Group | Biologic - Unite Biomatrix | Saline and Gauze
Number analyzed (Participants) | 42 | 48
Devices | 24 | 34

10. Secondary Outcome: Number of Device Removals
Description: Device removal is included in device failure under ITT. Subjects who experienced procedure-related events were also device failures under ITT. This endpoint is equivalent to device failure rates reported above.
Time Frame: Week 1 to Week 24
Population: ITT
Measure: Number; unit: Devices
Arm/Group | Biologic - Unite Biomatrix | Saline and Gauze
Number analyzed (Participants) | 42 | 48
Devices | 24 | 34

11. Secondary Outcome: Ease of Dressing Use
Description: Ease of usage on a 5-point scale where 1=greatest ease of use and 5=greatest difficult
Time Frame: Week 1 to Week 12
Population: ITT. Note: Limited information available since product no longer licensed with Baxter. The only stats analysis information available provides data for Unite Biomatrix treatment arm, and will need to assume analysis was not performed for control arm.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Biologic - Unite Biomatrix | Saline and Gauze
Number analyzed (Participants) | 42 | 0
Score on a Scale
  Ease of Preparation | 1.4 (0.6) |
  Handling | 1.2 (0.6) |
  Comfortability | 1.5 (0.7) |
  Securability | 1.4 (0.6) |

ADVERSE EVENTS:
Time Frame: Day -12 through Day 180
Description: Source vocabulary unknown.
Arm/Group | Biologic - Unite Biomatrix | Saline and Gauze
All-Cause Mortality (participants affected / at risk) | 1/42 | 2/48
Serious Adverse Events (participants affected / at risk) | 9/42 | 8/48
Other Adverse Events (participants affected / at risk) | 6/42 | 7/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biologic - Unite Biomatrix (N=42) | Saline and Gauze (N=48)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Infection (Infections and infestations) | 4 (4) | 2 (2)
Death (Investigations) | 1 (1) | 1 (1) — Cause of death unknown, arbitrarily selected body system of 'Investigations'
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Foot amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (General disorders) | 1 (1) | 0 (0)
Vomiting (General disorders) | 1 (1) | 0 (0)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biologic - Unite Biomatrix (N=42) | Saline and Gauze (N=48)
Infection (Infections and infestations) | 2 (3) | 3 (4)
Ulcer (Endocrine disorders) | 0 (0) | 2 (2)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Back Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study initially sponsored by Synovis Surgical Innovation, and product now licensed with Biomed Design. Unable to obtain all data for study. Clinical Study Report not located and results summarized from an abbreviated Statistical Analysis Report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days